CLINICAL TRIAL: NCT02182882
Title: Efficacy of Ginsana in Improving Half -Time Hemoglobin Re-oxygenation in Recreational Sportspeople: a Double Blind, Placebo Controlled Pilot Study
Brief Title: Efficacy of Ginsana in Improving Half-time Hemoglobin Re-oxygenation in Healthy People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1020.10
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- GINSANA (Experimental)
  Interventions: Drug: GINSANA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GINSANA
  Arms: GINSANA
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the efficacy of ginsana in improving half-time hemoglobin re-oxygenation in healthy, recreational sportspeople and to assess the safety of the product

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers between 18 and 40 years old
* Females must test negative for pregnancy
* Recreational athletes according to the american college of sports medicine (ACSM) definition
* Familiar with the cycle ergometer exercise methodology
* Written inform consent according to good clinical practice (GCP) and local regulations

Exclusion Criteria:

* Pre-treatment (less than 2 weeks prior to inclusion in this trial) and/or concomitant treatment with any drug that any drug that could have influence the trail methodology
* Alcohol and drug abuse (as defined in Diagnostic and Statistic Manual IV( DSM-IV)) per subject verbal report
* Smokers
* Known hypertension
* Known hypercholesterolemia (moderate/severe)
* Female volunteers taking oral or injectable contraceptives
* Female volunteers of child bearing potential not using adequate means of birth control, other than contraceptive pills [intrauterine devices (IUDs)]
* Pregnancy and/or lactation
* Liver and/or renal disease and/or vascular disease
* Relevant allergy or known hypersensitivity to the investigational drug or its excipients
* Participation in another clinical trial within the last 4 weeks and concurrent participation in another clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 1999-03; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in half-time hemoglobin re-oxygenation by Near InfraRed Spectroscopy (NIRS) methodology | Baseline, day 84 post first drug dispense

SECONDARY OUTCOMES:
Change from baseline in half-time hemoglobin re-oxygenation by NIRS methodology | Baseline, day 21, 42 and 63 post first drug dispense
Maximum endurance time | up to day 84 post first drug dispense
Change from baseline in respiratory threshold | Baseline, up to day 84 post first drug dispense
Change from baseline in thiobarbituric acid (TBARS) | Baseline, up to day 84 post first drug dispense
Change from baseline in glutathion superdismutase / glutathion superdismutase oxidised (GSA/GSSG) | Baseline, up to day 84 post first drug dispense